CLINICAL TRIAL: NCT05429983
Title: Assessing Stimulated Upper Airway Mechanics to Predict Outcomes in Hypoglossal Nerve
Brief Title: Predicting Outcomes in Hypoglossal Nerve Stimulation Therapy With Stimulated Upper Airway Mechanics
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: American Academy of Sleep Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00319723; 278-jf-22 (Other Grant/Funding Number: American Academy of Sleep Medicine)
Record Dates: First submitted 2022-06-17; First posted 2022-06-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypoglossal Nerve Stimulation Candidates: Participants will have a diagnosis of obstructive sleep apnea and have failed treatment with continuous positive airway pressure (CPAP). Participants will be those undergoing drug-induced sleep endoscopy (DISE) as part of routine clinical care for work up of hypoglossal nerve stimulation candidacy as a treatment for obstructive sleep apnea.

SUMMARY:
Obstructive sleep apnea (OSA) is a highly prevalent disease resulting from dynamic upper airway collapse during sleep. Continuous positive airway pressure (CPAP) is highly efficacious but high rates of non-adherence to CPAP leaves large number of OSA patients at risk for cardiometabolic sequelae. Inspire™ is an FDA-approved hypoglossal nerve stimulation device (HGNS) used in select patients with OSA who are intolerant of CPAP. The device consists of an implanted impulse generator with a stimulating cuff lead around the distal hypoglossal nerve. Despite these stringent selection criteria, up to one-third of patients implanted have inadequate responses to HGNS and remain at risk for complications from untreated OSA. The current proposal builds on routine clinical care to characterize upper airway biomechanics and determine predictors of clinical responses to HGNS therapy.

Drug induced sleep endoscopy (DISE) is a prerequisite for HGNS treatment and represents an ideal opportunity to rapidly characterize upper airway dynamics under controlled, standardized conditions. The amount of nasal pressure required to relieve airway obstruction (minimal therapeutic pressure) is a significant predictor of successful treatment of OSA with HGNS. As a result, CPAP titration (measuring pharyngeal collapse patterns at varying nasal pressures) has become an integral part of DISE to select parties for HGNS at multiple institutions. Nevertheless, changes in upper airway collapsibility in response HGNS may differ significantly between patients. This stud will examine if changes in upper airway patency with direct genioglossus muscle stimulation at the time of DISE predicts successful treatment with HGNS as defined by a 50% reduction on apnea-hypopnea index (AHI) and an on-treatment AHI <20.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants with moderate or severe sleep apnea (defined by > 15 apneas and hypopneas per hour of sleep), who are undergoing DISE as part of routine evaluation for Inspire hypoglossal nerve stimulation therapy or for ineffective HGNS therapy.

Exclusion Criteria:

* Significant cardiac disease, unstable or recent cardiac events
* Active pulmonary, liver or renal disease
* Uncontrolled hypertension (BP>160/100)
* Neuromuscular disease
* Major psychiatric disease
* Pregnancy
* Anticoagulation therapy (e.g. Coumadin, Dabigatran)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be those undergoing drug-induced sleep endoscopy as part of routine clinical care for work up hypoglossal nerve stimulation therapy candidacy. All participants will have a confirmed diagnosis of obstructive sleep apnea with an apnea-hypopnea index >15 and deemed to be intolerant of continuous positive airway pressure.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2027-11-29 (Estimated); Study Completion 2028-11-29 (Estimated)

PRIMARY OUTCOMES:
Tidal airflow with direct genioglossus stimulation | at the time of drug-induced sleep endoscopy, up to 1 hour
  Tidal airflow (mL) with direct stimulation of the genioglossus muscle will be measured at the time of drug-induced sleep endoscopy.
HGNS therapy success as assessed by the apnea hypopnea index | at 1 year post HGNS implantation
  Successful treatment with HGNS, as defined by a 50% reduction in apnea hypopnea index (AHI) and an on-therapy AHI of <15 (the same criteria as in major trials of non-CPAP OSA treatment).

SECONDARY OUTCOMES:
Therapeutic CPAP pressure with direct genioglossus stimulation | At the time of drug-induced sleep endoscopy, up to 1 hour
  Therapeutic CPAP pressure (cmH20) with direct stimulation of the genioglossus muscle will be measured at the time of drug-induced sleep endoscopy.
Airway critical closing pressure with direct genioglossus stimulation | At the time of drug-induced sleep endoscopy, up to 1 hour
  Airway critical closing pressure (cmH20) with direct stimulation of the genioglossus muscle will be measured at the time of drug-induced sleep endoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Motz, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No